CLINICAL TRIAL: NCT03135327
Title: Clinical Applications of Advanced Ophthalmic Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jianhua (Jay) Wang, MD, PhD, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20070492
Record Dates: First submitted 2017-04-24; First posted 2017-05-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Dry Eye Syndromes; Diabetic Retinopathy; Presbyopia; Myopia; Dementia
MeSH Terms: conditions — Multiple Sclerosis; Dry Eye Syndromes; Diabetic Retinopathy; Presbyopia; Myopia; Dementia | interventions — Ocufolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Phase - Ocufolin Group (Experimental): Participants in this group will receive the Ocufolin medical food for 6 months.
  Interventions: Dietary Supplement: Ocufolin
- Observational Phase Group (No Intervention): Participants in this group will be studied and followed up for 1-2 years.

INTERVENTIONS:
Dietary Supplement: Ocufolin — Ocufolin medical food capsules will be taken once a day by mouth each morning with a meal for the first week, two capsules orally each morning with a meal for the second week and three capsules orally each morning with a meal for the rest of the 6 months study duration.
  Arms: Interventional Phase - Ocufolin Group

SUMMARY:
The purpose of this study is to determine the clinical application of advanced ophthalmic imaging devices such as optical coherence tomography (OCT), retinal function imager (RFI), slit-lamp biomicroscopy (SLB), PERG in diseased eyes and normal controls.

There are two phases in this study. The first phase is an observational phase which studies the eye in various conditions. The second phase is an interventional phase which studies the changes in the eyes after taking an over-the-counter medical food (Ocufolin) for 6 months.

ELIGIBILITY:
Observational Phase 1 Group

Inclusion Criteria:

1. Self-reported normal healthy subjects;
2. Clinical diagnosis of Alzheimer's Disease, mild cognitive impairment, multiple sclerosis, dry eye, myopia, diabetics and stroke;
3. Who can keep the eye open for imaging.

Exclusion Criteria:

1. who can not read and sign the ICF;
2. who can not receiving ophthalmic imaging;
3. who cannot tolerate bright light during imaging.

Interventional Phase 2 Group:

Inclusion criteria

The participant will be eligible for entry in the study if s/he:

1. Is at least 18 years old and has full legal capacity to volunteer;
2. Has read and signed the IRB Informed Consent Document;
3. Is willing and able to follow participant instructions;
4. Has clear corneas and crystalline lens;
5. Initial visual acuities were 20/80 or better;
6. MTHFR C677TT homozygous, or MTHFR C677T/A1298C compound heterozygous with mild to moderate micro-aneurismal vascular retinopathy disease;
7. Hemoglobin A1c is 10 or less;
8. Normotensive with or without medications;
9. Without retinal capillary dropout or macular edema;
10. Blood homocysteine > 9.

Exclusion criteria

The subjects will be ineligible for entry into the study if s/he:

1. Has an active ocular disease;
2. Has had surgery or an eye injury within 6 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Retinal microstructure using OCT. | up to 2 years
  Optical coherence tomography is used to measure the thickness of intraretinal layers. The measurement is in micrometer.
Retinal vasculature by optical coherence tomography angiography (OCTA) | up to 2 years
  Retinal vascular network density in percentage.
Conjunctival vasculature by functional slit-lamp (FSLB) | up to 2 years
  Conjunctival vascular network density in percentage.
Corneal epithelial thickness | up to 2 years
  Measured in micrometers using ultra high resolution OCT
Tear film thickness | up to 2 years
  Measured in micrometers using ultra high resolution OCT

SECONDARY OUTCOMES:
Retinal blood flow velocity by retinal function imager (RFI) | up to 2 years
  Retinal blood flow velocity in mm/s
Conjunctival blood flow velocity by functional slit-lamp (FSLB) | up to 2 years
  Conjunctival blood flow velocity in mm/s

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wang, MD, PhD, Principal Investigator — Bascom Palmer Eye Institute, University of Miami, Miami, FL
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No